CLINICAL TRIAL: NCT00617669
Title: A Phase III, Randomised, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of 10 mg ZD4054 (Zibotentan) in Combination With Docetaxel in Comparison With Docetaxel in Patients With Metastatic Hormone-resistant Prostate Cancer
Brief Title: A Phase III Trial of ZD4054 (Zibotentan) (Endothelin A Antagonist) and Docetaxel in Metastatic Hormone Resistant Prostate Cancer
Acronym: ENTHUSE M1C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4320C00033
Record Dates: First submitted 2008-01-24; First posted 2008-02-18 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: Hormone Resistant Prostate Cancer; Endothelin A Receptor Antagonist; Endothelin A; Endothelin A antagonist
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; ZD4054

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo + Docetaxel (Active Comparator): placebo oral tablet once daily + docetaxel intravenous infusion every 3 weeks
  Interventions: Drug: Docetaxel; Drug: Placebo
- ZD4054 + Docetaxel (Experimental): ZD4054 10 mg oral tablet once daily + docetaxel intravenous infusion every 3 weeks
  Interventions: Drug: Docetaxel; Drug: ZD4054

INTERVENTIONS:
Drug: Docetaxel — intravenous infusion given every three weeks
  Other Names: Taxotere®
Drug: ZD4054 — 10 mg oral once daily dose
  Other Names: Zibotentan
  Arms: ZD4054 + Docetaxel
Drug: Placebo — placebo oral tablet once daily
  Arms: Placebo + Docetaxel

SUMMARY:
Enthuse M1C is a large phase III clinical trial studying the safety and efficacy of ZD4054 (Zibotentan) in combination with docetaxel (Taxotere) in patients with metastatic hormone resistant prostate cancer (HRPC).

This clinical trial will test if the Endothelin A Receptor Antagonist ZD4054 (Zibotentan) can further improve survival compared with docetaxel alone.

ZD4054 (Zibotentan) is a new type of agent, which is thought to slow tumour growth and spread by blocking Endothelin A receptor activity. This trial will look at the effects of ZD4054 (Zibotentan) in hormone resistant prostate cancer patients with bone metastases compared with docetaxel.

All patients participating in this clinical trial will receive docetaxel chemotherapy, which is a commonly used chemotherapy to treat prostate cancer in addition to other existing prostate cancer therapies.

Half the patients will receive ZD4054 (Zibotentan), and half the patients will receive placebo in addition to docetaxel and other prostate cancer therapy. By participating in this trial there is a 50% chance that patients will receive an agent that may further slow the progression of the tumour.

No patients will be deprived of standard prostate cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients who answer TRUE to the following criteria may be eligible to participate in this trial.

* Confirmed diagnosis of prostate cancer (adenocarcinoma of the prostate) that has spread to the bone (bone metastasis)
* Increasing Prostate Specific Antigen (PSA), collected within one year of enrollment
* Currently receiving treatment with surgical or medical castration

Exclusion Criteria:

Patients who answer TRUE to the following ARE NOT eligible to participate in this trial.

* Previous treatment with chemotherapy (paclitaxel, docetaxel, and mitoxantrone). Prior targeted cancer therapies are permitted if received during a previous clinical trial.
* Suffering from heart failure or had a myocardial infarction within last 6 months
* A history of epilepsy or seizures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1494 (Actual)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Judd W Moul, MD, FACS, Principal Investigator — Duke University
Locations (147):
- United States (25):
  - Research Site, Greenbrae, California
  - Research Site, San Diego, California
  - Research Site, Norwich, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Ocala, Florida
  - Research Site, PORTUGALt Saint Lucie, Florida
  - Research Site, Rockville, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (3):
  - Research Site, Bahía Blanca, Buenos Aires
  - Research Site, Buenos Aires, Buenos Aires
  - Research Site, Santa Fe, Santa Fe Province
- Australia (9):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Redcliffe, Queensland
  - Research Site, Ashford, South Australia
  - Research Site, Footscray, Victoria
  - Research Site, Wodonga, Victoria
  - Research Site, Perth, Western Australia
  - Research Site, Subiaco, Western Australia
- Brazil (11):
  - Research Site, Fortaleza, Ceara/ LA
  - Research Site, Goiânia, Goias/ LA
  - Research Site, Goiânia, Goiás
  - Research Site, Belo Horizonte, Minas GERMANYais
  - Research Site, Curitiba, Parana/ Brazil
  - Research Site, Londrina, Paraná
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, PORTUGALto Alegre, Rio Grande Do Sul/ LA
  - Research Site, Ribeirão Preto, Sao Paulo/ LA
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
- Canada (6):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Czechia (7):
  - Research Site, Olomouc, Czech Republic
  - Research Site, Prague, Czech Republic
  - Research Site, Ústí nad Labem, Czech Republic
  - Research Site, Brno, Czechoslovakia Republic
  - Research Site, Jablonec nad Nisou
  - Research Site, Kroměříž
  - Research Site, Prague
- Finland (3):
  - Research Site, Helsinki, Finland
  - Research Site, Joensuu
  - Research Site, Seinäjoki
- France (8):
  - Research Site, La Roche-sur-Yon, FRANCEnce
  - Research Site, Marseille, FRANCEnce
  - Research Site, Paris, FRANCEnce
  - Research Site, Reims, FRANCEnce
  - Research Site, Villejuif, FRANCEnce
  - Research Site, Paris, Paris
  - Research Site, Saint-Herblain, Saint Herblain
  - Research Site, Paris
- Germany (11):
  - Research Site, Hanover, GERMANYmany
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Dresden
  - Research Site, Emmendingen
  - Research Site, Kirchheim-Teck
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Münster
  - Research Site, Tübingen
  - Research Site, Wuppertal
- Hungary (5):
  - Research Site, Budapest, HUNGARYary
  - Research Site, Győr, HUNGARYary
  - Research Site, Miskolc, HUNGARYary
  - Research Site, Ny Regyh Za, HUNGARYary
  - Research Site, Szeged, HUNGARYary
- India (11):
  - Research Site, Bangalore, Karnataka
  - Research Site, Trivandrum, Kerala
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Pune, Maharashtra
  - Research Site, Bikaner, Rajasthan
  - Research Site, Jaipur, Rajasthan
  - Research Site, Vellore, Tamil Nadu
  - Research Site, Kolkata, West Bengal
  - Research Site, Kolkota, West Bengal
  - Research Site, Delhi
  - Research Site, New Delhi
- Italy (3):
  - Research Site, Genoa, Italy
  - Research Site, Lugo (RA), Italy
  - Research Site, Rome, Italy
- Research Site, Nijmegen, Netherlands
- Peru (4):
  - Research Site, Cercado de Arequipa, Arequipa
  - Research Site, Cercado, Arequipa
  - Research Site, Callao
  - Research Site, Lima
- Poland (5):
  - Research Site, Lublin, POLANDand
  - Research Site, Swidnica, POLANDand
  - Research Site, Warszaa, POLANDand
  - Research Site, Kościerzyna
  - Research Site, Wroclaw
- Portugal (2):
  - Research Site, Coimbra, PORTUGALtugal
  - Research Site, PORTUGALto, PORTUGALtugal
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Sibiu
  - Research Site, Timișoara
- Russia (5):
  - Research Site, Barnaul, RUSSIAsia
  - Research Site, Izhevsk, RUSSIAsia
  - Research Site, Kursk, RUSSIAsia
  - Research Site, Sochi, RUSSIAsia
  - Research Site, Voronezh, RUSSIAsia
- Serbia (2):
  - Research Site, Belgrade, SERBIAbia
  - Research Site, Niš, SERBIAbia
- South Africa (5):
  - Research Site, Panorama, Cape Town
  - Research Site, TyGERberg, Cape Town
  - Research Site, Overport, Durban
  - Research Site, Bloemfontein
  - Research Site, Port Elizabeth
- South Korea (5):
  - Research Site, Ilsandong-gu, Goyang-si, Gyeonggi-do
  - Research Site, Cheongju-si, North Chungcheong
  - Research Site, Nowon-gu, Seoul
  - Research Site, Seodaemun-gu, Seoul
  - Research Site, Songpa-gu, Seoul
- Spain (2):
  - Research Site, Madrid, Spain
  - Research Site, Valencia, Spain
- Sweden (2):
  - Research Site, Stockholm, Sweden
  - Research Site, Uppsala
- Switzerland (3):
  - Research Site, Aarau
  - Research Site, Locarno
  - Research Site, Sursee
- Taiwan (2):
  - Research Site, Kaohsiung City, TAIWANwan
  - Research Site, TAIWANpei, TAIWANwan
- United Kingdom (4):
  - Research Site, Reading, Berkshire
  - Research Site, Manchester, Manchester
  - Research Site, Westgate Road, Newcastle Upon Tyne
  - Research Site, London

REFERENCES:
- [Derived] Fizazi K, Higano CS, Nelson JB, Gleave M, Miller K, Morris T, Nathan FE, McIntosh S, Pemberton K, Moul JW. Phase III, randomized, placebo-controlled study of docetaxel in combination with zibotentan in patients with metastatic castration-resistant prostate cancer. J Clin Oncol. 2013 May 10;31(14):1740-7. doi: 10.1200/JCO.2012.46.4149. Epub 2013 Apr 8. PMID 23569308

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1494 patients with hormone resistant prostate cancer patients and bone metastasis were recruited between 24th January 2008 and 10th May 2011
Pre-assignment Details: 442 of the 1494 enrolled patients were not randomised to treatment groups as they failed screening.
Groups:
- ZD4054 + Docetaxel: XD4054 10 mg oral tablet once daily + docetaxel intravenous infusion every 3 weeks
Period: Overall Study
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Started | 524 | 528
Patients Who Received IP | 522 | 525
Completed | 94 (Patients receiving ZD4054 10 mg at data cut-off) | 77 (Patients receiving placebo at data cut-off)
Not Completed | 430 | 451
Not completed — Withdrawal by Subject | 71 | 77
Not completed — Lost to Follow-up | 3 | 2
Not completed — Adverse Event | 87 | 76
Not completed — Protocol Violation | 2 | 3
Not completed — Reason not otherwise captured, eg; death | 265 | 290
Not completed — Patients randomized but not treated | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 524 | 528 | 1052
Age Continuous [Mean (Standard Deviation); unit: years]
  overall | 8.1 (67.7) | 7.8 (67.6) | 7.9 (67.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 524 | 528 | 1052

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Median time (in months) from randomisation until death using the Kaplan-Meier method.
Time Frame: Patients were followed for survival up to 40 months
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 524 | 528
Months | 20.0 [11.6 to 32.0] | 19.2 [12.0 to 30.3]

2. Secondary Outcome: Progression Free Survival
Description: Median time (in months) from randomisation until clinical progression of disease using the Kaplan-Meier method. Progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline
Time Frame: Patients were followed for progression up to 40 months
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 524 | 528
Months | 7.0 [3.5 to 13.1] | 7.9 [4.0 to 12.6]

3. Secondary Outcome: Incidence of Skeletal Related Events
Description: Median time (in months) from randomisation until occurrence of a skeletal related event using the Kaplan-Meier method, where skeletal related event is defined as the first occurrence of a pathological fracture, a vertebral compression fracture not related to trauma, prophylactic surgery or radiation for impending fracture or spinal cord compression, or a spinal cord compression.
Time Frame: While receiving docetaxel study visits were aligned with its administration ie every 3weeks, after 12 weeks and completion of docetaxel therapy every 12 weeks (up to 40 months)
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 524 | 528
Months | 17.4 [10.0 to 25.3] | 17.3 [10.3 to 26.0]

4. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Median time (in months) from randomisation until first PSA value >50% higher than baseline of at least 5ng/ml seen in at least 2 consecutive PSA values at least 2 weeks apart using the Kaplan-Meier method.
Time Frame: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 524 | 528
Months | 11.9 [6.2 to 19.6] | 12.1 [6.0 to 18.3]

5. Secondary Outcome: Time to Pain Progression
Description: Median time (in months) from randomisation until date of first assessment of increased pain using the Kaplan-Meier method, where increased pain event is defined as the first of a patient requiring opiate medication for duration of ≥1 week for pain due to prostate cancer metastasis, pain due to metastasis that has an increase in the worst pain item of the Brief Pain Inventory (BPI) from baseline to a minimum score of 5 with no decrease in analgesic use, or pain due to metastasis requiring radionuclide therapy, radiation therapy or surgery.
Time Frame: as for outcome 3
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 524 | 528
Months | 9.3 [3.9 to 18.4] | 10.0 [4.2 to 18.6]

6. Secondary Outcome: Pain Response
Description: Number of patients with a pain response, defined as a decrease in brief pain inventory questionnaire (BPI) of at least 2 points from baseline or a decrease in opiate use of 25% from baseline.
Time Frame: as for outcome 3
Population: The Pain Response Analysis Set includes patients who were either receiving opiates at baseline (randomisation) or with a baseline BPI score ≥2.
Measure: Number; unit: Participants
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 362 | 373
Participants | 255 | 276

7. Secondary Outcome: Health Related Quality of Life
Description: Median time (in months) from randomisation until deterioration of Health Related Quality of Life using the Kaplan-Meier method, where deterioration is defined as a change from baseline of less than or equal to -6 points in Total FACT-P score maintained for 2 consecutive visits.
Time Frame: as for outcome 3
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 524 | 528
Months | 4.4 [1.6 to 10.7] | 5.1 [2.1 to 12.0]

8. Secondary Outcome: PSA Response
Description: PSA response defined as >50% decrease in serum PSA values from baseline seen in at least 2 consecutive PSA values at least 2 weeks apart.
Time Frame: as for outcome 3
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 524 | 528
Participants | 279 | 298

ADVERSE EVENTS:
Arm/Group | ZD4054 + Docetaxel | Placebo + Docetaxel
Serious Adverse Events (participants affected / at risk) | 214/522 | 203/525
Other Adverse Events (participants affected / at risk) | 490/522 | 483/525
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054 + Docetaxel (N=522) | Placebo + Docetaxel (N=525)
Febrile Neutropenia (Blood and lymphatic system disorders) | 22 | 16
Anaemia (Blood and lymphatic system disorders) | 19 | 8
Neutropenia (Blood and lymphatic system disorders) | 10 | 12
Leukopenia (Blood and lymphatic system disorders) | 2 | 4
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphatic Obstruction (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 5 | 2
Cardiac Failure (Cardiac disorders) | 5 | 2
Acute Myocardial Infarction (Cardiac disorders) | 3 | 4
Angina Pectoris (Cardiac disorders) | 2 | 2
Atrial Flutter (Cardiac disorders) | 1 | 2
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 2
Coronary Artery Stenosis (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 2
Myocardial Ischaemia (Cardiac disorders) | 0 | 2
Ventricular Tachycardia (Cardiac disorders) | 0 | 2
Angina Unstable (Cardiac disorders) | 0 | 1
Aortic Valve Disease (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 1
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Diastolic Dysfunction (Cardiac disorders) | 0 | 1
Hypertrophic Cardiomyopathy (Cardiac disorders) | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 1 | 0
Adrenocortical Insufficiency Acute (Endocrine disorders) | 0 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Scleral Disorder (Eye disorders) | 1 | 0
Staphyloma (Eye disorders) | 0 | 1
Visual Acuity Reduced (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Constipation (Gastrointestinal disorders) | 3 | 3
Ileus (Gastrointestinal disorders) | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Anal Fistula (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0
Colonic Polyp (Gastrointestinal disorders) | 1 | 0
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 1
Erosive Oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 0 | 1
Intestinal Infarction (Gastrointestinal disorders) | 1 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0
Neutropenic Colitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectourethral Fistula (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 6 | 12
Death (General disorders) | 10 | 6
Oedema Peripheral (General disorders) | 6 | 3
General Physical Health Deterioration (General disorders) | 0 | 3
Asthenia (General disorders) | 0 | 2
Disease Progression (General disorders) | 1 | 2
Medical Device Complication (General disorders) | 0 | 2
Chest Pain (General disorders) | 1 | 0
Device Occlusion (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Pneumonia (Infections and infestations) | 26 | 8
Sepsis (Infections and infestations) | 10 | 2
Urinary Tract Infection (Infections and infestations) | 9 | 7
Urosepsis (Infections and infestations) | 4 | 5
Cellulitis (Infections and infestations) | 4 | 1
Neutropenic Sepsis (Infections and infestations) | 4 | 3
Bronchopneumonia (Infections and infestations) | 3 | 2
Lung Infection (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 2
Infection (Infections and infestations) | 0 | 2
Lobar Pneumonia (Infections and infestations) | 0 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 2
Pharyngitis (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0
Skin Infection (Infections and infestations) | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Arthritis Bacterial (Infections and infestations) | 0 | 1
Arthritis Infective (Infections and infestations) | 0 | 1
Bacterial Diarrhoea (Infections and infestations) | 1 | 0
Catheter Site Infection (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 0 | 1
Lyme Disease (Infections and infestations) | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 1 | 0
Neutropenic Infection (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 1 | 0
Peritonitis Bacterial (Infections and infestations) | 1 | 0
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 1
Psoas Abscess (Infections and infestations) | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 2
Cerebral Haemorrhage Traumatic (Injury, poisoning and procedural complications) | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1
Kidney Rupture (Injury, poisoning and procedural complications) | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 | 1
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Stress Fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 2 | 0
Blood Electrolytes Abnormal (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT Prolonged (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil Count Decreased (Injury, poisoning and procedural complications) | 0 | 1
Transaminases Increased (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 7 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 2 | 2
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo Maligna Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Lymphoid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 3 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 2
Cerebral Infarction (Nervous system disorders) | 1 | 2
Presyncope (Nervous system disorders) | 1 | 2
Transient Ischaemic Attack (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 0 | 1
Depressed Level Of Consciousness (Nervous system disorders) | 1 | 0
Diabetic Neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Completed Suicide (Psychiatric disorders) | 1 | 3
Confusional State (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 7 | 2
Haematuria (Renal and urinary disorders) | 2 | 4
Urinary Retention (Renal and urinary disorders) | 1 | 2
Bladder Neck Obstruction (Renal and urinary disorders) | 1 | 0
Bladder Obstruction (Renal and urinary disorders) | 1 | 0
Calculus Ureteric (Renal and urinary disorders) | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Cystitis Noninfective (Renal and urinary disorders) | 0 | 1
Haemorrhage Urinary Tract (Renal and urinary disorders) | 1 | 0
Postrenal Failure (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Tubular Necrosis (Renal and urinary disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 3 | 2
Aortic Aneurysm (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 2
Jugular Vein Thrombosis (Vascular disorders) | 0 | 2
Circulatory Collapse (Vascular disorders) | 0 | 1
Femoral Artery Occlusion (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypovolaemic Shock (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 1 | 0
sThrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054 + Docetaxel (N=522) | Placebo + Docetaxel (N=525)
Anaemia (Blood and lymphatic system disorders) | 155 | 116
Neutropenia (Blood and lymphatic system disorders) | 114 | 118
Leukopenia (Blood and lymphatic system disorders) | 64 | 60
Lacrimation Increased (Eye disorders) | 38 | 36
Diarrhoea (Gastrointestinal disorders) | 183 | 185
Nausea (Gastrointestinal disorders) | 174 | 160
Constipation (Gastrointestinal disorders) | 152 | 129
Vomiting (Gastrointestinal disorders) | 110 | 84
Dyspepsia (Gastrointestinal disorders) | 21 | 40
Stomatitis (Gastrointestinal disorders) | 32 | 35
Abdominal Pain (Gastrointestinal disorders) | 25 | 34
Abdominal Pain Upper (Gastrointestinal disorders) | 31 | 27
Oedema Peripheral (General disorders) | 278 | 188
Fatigue (General disorders) | 150 | 164
Asthenia (General disorders) | 118 | 117
Pyrexia (General disorders) | 59 | 60
Mucosal Inflammation (General disorders) | 37 | 28
Rhinitis (Infections and infestations) | 51 | 36
Urinary Tract Infection (Infections and infestations) | 37 | 48
Nasopharyngitis (Infections and infestations) | 30 | 36
Upper Respiratory Tract Infection (Infections and infestations) | 18 | 27
Weight Decreased (Infections and infestations) | 37 | 37
Decreased Appetite (Metabolism and nutrition disorders) | 127 | 119
Hypocalcaemia (Metabolism and nutrition disorders) | 29 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 27
Back Pain (Musculoskeletal and connective tissue disorders) | 94 | 91
Arthralgia (Musculoskeletal and connective tissue disorders) | 80 | 86
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 71 | 84
Myalgia (Musculoskeletal and connective tissue disorders) | 42 | 53
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 46 | 28
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 22 | 37
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 29 | 37
Bone Pain (Musculoskeletal and connective tissue disorders) | 28 | 32
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 32 | 20
Headache (Nervous system disorders) | 107 | 71
Dysgeusia (Nervous system disorders) | 88 | 73
Neuropathy Peripheral (Nervous system disorders) | 49 | 65
Paraesthesia (Nervous system disorders) | 45 | 48
Dizziness (Nervous system disorders) | 43 | 45
Peripheral Sensory Neuropathy (Nervous system disorders) | 41 | 39
Hypoaesthesia (Nervous system disorders) | 24 | 28
Insomnia (Psychiatric disorders) | 71 | 59
Haematuria (Renal and urinary disorders) | 30 | 17
Dysuria (Renal and urinary disorders) | 29 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 82 | 72
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 78
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 78 | 26
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 43 | 38
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 | 31
Alopecia (Skin and subcutaneous tissue disorders) | 178 | 196
Rash (Skin and subcutaneous tissue disorders) | 24 | 40
Nail Discolouration (Skin and subcutaneous tissue disorders) | 28 | 39
Dry Skin (Skin and subcutaneous tissue disorders) | 32 | 28
Nail Disorder (Skin and subcutaneous tissue disorders) | 23 | 28
Hypertension (Vascular disorders) | 16 | 37
Hypotension (Vascular disorders) | 33 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
3. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

AstraZeneca can review results communications prior to public release and may within 60 days of receipt require amendments to be made. AstraZeneca can also require that submission or disclosure be delayed to allow for